CLINICAL TRIAL: NCT02327754
Title: Effect of Topiroxostat on Urinary Albumin Excretion in Patients With eARly Stage Diabetic Nephropathy and Hyperuricemia With or Without Gout: a Randomized, Placebo-controlled, Double-blind Phase 2a Trial (UPWARD).
Brief Title: Effect of Topiroxostat on Urinary Albumin Excretion Early Stage Diabetic Nephropathy and Hyperuricemia With or Without Gout
Acronym: UPWARD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FY1004
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-11

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active comparator (Active Comparator): Topiroxostat, (Oral daily dosing for 28 weeks)
  Interventions: Drug: Topiroxostat BID, (Oral daily dosing for 28 weeks)
- Placebo comparator (Placebo Comparator): Placebo, (Oral daily dosing for 28 weeks)
  Interventions: Drug: Placebo BID, (Oral daily dosing for 28 weeks)

INTERVENTIONS:
Drug: Topiroxostat BID, (Oral daily dosing for 28 weeks) — The dose of topiroxostat is increased up to 160 mg/day in a stepwise manner.
  Arms: Active comparator
Drug: Placebo BID, (Oral daily dosing for 28 weeks) — Subjects randomized to the placebo arm will receive placebo.
  Arms: Placebo comparator

SUMMARY:
The purpose of this study is to investigate the effect of topiroxostat on urinary albumin excretion and the safety in patients with early stage diabetic nephropathy and hyperuricemia with or without gout. Participants are randomized to placebo (n=20) or topiroxostat (n=40) for 28 weeks. The investigational drugs for this study are supplied by FUJI YAKUHIN CO., LTD.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes patients
* Clinically or pathologically diagnosed diabetic nephropathy
* Hyperuricemic or gout patients
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/1.73m^2 and urine albumin creatinine ratio (UACR) greater than or equal to 45 and less than 300 mg/g

Exclusion Criteria:

* Patient has known non-diabetic nephropathy (other than nephrosclerosis)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine albumin creatinine ratio | 28 weeks

SECONDARY OUTCOMES:
sUA, eGFR, L-FABP, HbA1c, SBP, DBP, TC | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sanwa Kagaku Kenkyusho Co., Ltd., Nagoya, Aichi-ken, Japan